CLINICAL TRIAL: NCT02305043
Title: Identification of Biomarkers for Prediction of Response or Resistance Against Target Therapy in Adenocarcinoma of the Stomach or Gastroesophageal Junction. A Non-interventional Study
Brief Title: Identification of Biomarkers for Prediction of Response or Resistance Against Target Therapy in Gastric Cancer
Acronym: VARIANZ
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Florian Lordick, MD, Director University Cancer Center Leipzig, University of Leipzig
Other Study IDs: VARIANZ; 01ZX1310E (Other Grant/Funding Number: Federal Ministry of Education and Research)
Record Dates: First submitted 2014-11-17; First posted 2014-12-02 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms
Keywords: non-interventional; advanced gastric cancer; Trastuzumab; HER2
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: non-interventional — non-interventional

SUMMARY:
The aim of this study is to identify biomarkers predicting response or resistance factors of a targeted therapy with trastuzumab in advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven adenocarcinoma of the stomach or gastroesophageal junction

  * stage IV
  * patient receives chemotherapy
  * signed informed consent
  * Age > 18 years

Exclusion Criteria:

* Patient can not understand meaning and purpose of the study
* patient already received a chemotherapy treatment for advanced disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffer from histologically proven adenocarcinoma of the stomach or gastroesophageal junction
Sampling Method: Non-Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2014-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Objective Response | 12 months
  Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR). CR is defined as the disappearance of all target lesions. PR is defined as at least 30% decrease in the sum of the longest dimension of the target lesion

SECONDARY OUTCOMES:
time-to-progression | up to 24 months
  The period from study entry until disease progression, death, or date of last contact.
overall survival | up to 24 months
  OS is the duration from enrollment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, Prof., Principal Investigator — University Cancer Center Leipzig
Locations (1):
- University Cancer Center Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Wang J, Sun N, Kunzke T, Shen J, Feuchtinger A, Wang Q, Meixner R, Gleut RL, Haffner I, Luber B, Lordick F, Walch A. Metabolic heterogeneity affects trastuzumab response and survival in HER2-positive advanced gastric cancer. Br J Cancer. 2024 Apr;130(6):1036-1045. doi: 10.1038/s41416-023-02559-6. Epub 2024 Jan 24. PMID 38267634
- [Derived] Ebert K, Haffner I, Zwingenberger G, Keller S, Raimundez E, Geffers R, Wirtz R, Barbaria E, Hollerieth V, Arnold R, Walch A, Hasenauer J, Maier D, Lordick F, Luber B. Combining gene expression analysis of gastric cancer cell lines and tumor specimens to identify biomarkers for anti-HER therapies-the role of HAS2, SHB and HBEGF. BMC Cancer. 2022 Mar 9;22(1):254. doi: 10.1186/s12885-022-09335-4. PMID 35264144
- [Derived] Haffner I, Schierle K, Raimundez E, Geier B, Maier D, Hasenauer J, Luber B, Walch A, Kolbe K, Riera Knorrenschild J, Kretzschmar A, Rau B, Fischer von Weikersthal L, Ahlborn M, Siegler G, Fuxius S, Decker T, Wittekind C, Lordick F. HER2 Expression, Test Deviations, and Their Impact on Survival in Metastatic Gastric Cancer: Results From the Prospective Multicenter VARIANZ Study. J Clin Oncol. 2021 May 1;39(13):1468-1478. doi: 10.1200/JCO.20.02761. Epub 2021 Mar 25. PMID 33764808